CLINICAL TRIAL: NCT06815263
Title: Listener Training for Improved Intelligibility of People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14004; 1R01DC020930 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Dysarthria, Hypokinetic
Keywords: Dysarthria; Parkinson's disease; Speech; Listener
MeSH Terms: conditions — Dysarthria; Speech

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Condition (Experimental): Listener receives speech of patient with dysarthria
  Interventions: Behavioral: Listener Training
- Control condition (Sham Comparator): Listener receives speech of speaker with no speech disorder
  Interventions: Behavioral: Listener Training

INTERVENTIONS:
Behavioral: Listener Training — Partner participants are presented with individual audio phrases that make up passage reading speech stimuli and orthographic transcriptions of what the patient is saying. Partners are asked to listen carefully to the audio files and use the written subtitles to help them understand what is being said.

SUMMARY:
Listener training offers a promising avenue for improving communication for people with dysarthria due to Parkinson's disease by offsetting the intelligibility burden from the patient onto their primary communication partners. Here, we employ a repeated-measures, randomized controlled trial to establish the efficacy of listener training for patients with PD and their primary communication partners. This translational work will establish a new realm of clinical practice in which the intelligibility impairments in PD are addressed by training partners to better understand dysarthric speech, thus elevating communication outcomes and participation in daily life.

DETAILED DESCRIPTION:
People with dysarthria due to Parkinson's disease (PD) frequently present with reduced intelligibility, which can have significant consequences, including reduced participation in situations involving communicating with others and resulting in social isolation.1-5 Few effective treatments exist to ease the intelligibility burden of dysarthria in PD, and most require significant cognitive and physical effort on the part of the speaker to achieve and maintain gains.6,7 Once people with PD have progressed beyond the early stages of the disease, and their cognitive and physical impairments limit their ability to use traditional speech therapy techniques, they are not realistic treatment candidates for current interventions; and no other interventions are available to support their communication. This is a serious and consequential gap in clinical care for people with PD. The current proposal addresses this critical gap by shifting the weight of behavioral change from the speaker to the listener, specifically key communication partners such as family. Indeed, for older adults, most of their time spent with others is spent with family members.8 Further, key partners of patients with PD wish to have a more significant and active role in communication rehabilitation.9,10 A listener-targeted remediation approach for intelligibility impairments in people with dysarthria and PD is firmly grounded in theoretical models of perceptual learning11-13 and rigorously supported by our decade-long research program targeting perceptual learning of dysarthric speech.14-30 To date, this line of investigation has chiefly targeted the theory of listener adaptation to the degraded signal; however, robust intelligibility improvements of up to 20 percent across studies have been observed.15 With a rigorous account of how and what listeners adapt to, we are ideally positioned to move this work from bench to bedside, establishing listener (i.e., perceptual) training as a clinical intervention to improve intelligibility in people with PD. Here, we establish the efficacy of listener training for patients with PD and their primary communication partners using a repeated-measures, randomized controlled trial (SA1). Immediate acquisition and retention of intelligibility improvements will be examined as a function of speaker severity. We then evaluate three theoretically and empirically-motivated communication benefits of listener training that extend beyond intelligibility, including listening effort, comprehension, and communicative participation (SA2). Finally, we engage stakeholder input to inform clinical implementation of listener training using qualitative semi-structured interviews (SA3) with patients with PD and their partners. This will provide insights into the effectiveness and feasibility of the intervention approach, ensuring that their needs and preferences are considered and that they feel empowered and motivated for a listener training approach. Thus, in three independent aims, this proposal will address a current void in our clinical toolbox, establishing a new realm of clinical practice in which communication challenges in PD are managed by training partners to better understand the degraded speech.

ELIGIBILITY:
Inclusion Criteria:

* Primary language is English
* 18 years or older
* medical diagnosis of Parkinson's disease (patient participants)
* speech diagnosis of hyperkinetic dysarthria, exhibiting hallmark characteristics (patient participants)

Exclusion Criteria:

* Severe cognitive impairment
* Less than 18 years of age
* Primary language other than English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-03-26 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Speech intelligibility | pretest, during training, immediate posttest, one week posttest, one month posttest
  Percent words correct (PWC)

SECONDARY OUTCOMES:
Listening effort | Pretest, one week posttest, one month posttest
  Rating scale, 0-100 scale with question "how easy is this speech to understand", with endpoints of 'difficult' on the zero side and 'easy' on the 100 side
Comprehension | Pretest, one week posttest, one month posttest
  Story comprehension accuracy score, listeners answer a series of multiple choice comprehension questions, accuracy is defined as how many correct responses they choose for each story
Communicative Participation Item Bank | Pretest, one month posttest
  Patient and partner reported summed score across different communication situations

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Borrie, PhD, Principal Investigator — Utah State University; Kaitlin Lansford, PhD, Principal Investigator — Florida State University; Sarah Yoho Leopold, PhD, Study Director — Utah State University
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Utah State University, Logan, Utah

IPD SHARING:
Plan to Share IPD: Undecided